CLINICAL TRIAL: NCT03859453
Title: Follow-up in Early and Locally Advanced Breast Cancer Patients
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: European Organisation for Research and Treatment of Cancer - EORTC (Network)
Responsible Party: Sponsor
Other Study IDs: EORTC-1617-QLG-BCG
Record Dates: First submitted 2019-02-28; First posted 2019-03-01 (Actual); Last update posted 2024-01-24 (Actual); Status verified 2024-01

CONDITIONS: Breast Cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
A cross-sectional follow-up study of Early and Locally Advanced Breast Cancer patients after primary treatment.

DETAILED DESCRIPTION:
The objective of this study is to assess follow-up patterns and identify patients with increased levels of physical and/or psychosocial problems after treatment in early breast cancer and locally advanced breast cancer.

830 patients stratified by cancer sites and treatment - a minimum of 120 patients within each stratum - will be recruited.

Institutional data on follow-up policy, demographic and clinical data (related to treatment history and tumor characteristics) will be collected. Patients will complete a set of 139 Quality of Life questions, at one single time point.

Statistical analysis includes descriptive statistic for socio-demographic and clinical data, overall and per treatment, age and risk group. Patterns of follow-up will be identified and described overall, and per treatment, age, risk group and country.

Where available, normative data will be used to identify those QoL domains where there is a clinically relevant difference with the general population.

Multivariable model building will be used to build predictive models on the overall population to investigate determinants for the physical, sexual and emotional needs based on the identified PROM outcomes. Factor analysis will be undertaken to investigate the inter-correlations between physical, sexual and emotional needs in the overall population and in the relevant subgroups of interest.

The magnitude of the observed differences will be assessed by clinical important effect size rather than by statistical significance.

ELIGIBILITY:
Inclusion Criteria:

* Histologically proven Early Breast Cancer (EBC) and Locally Advanced Breast Cancer (LABC) patients who have completed their primary treatment (except endocrine therapy), between 12 months and 36 months after the diagnosis.
* Disease-free without any evidence of relapse
* Age ≥ 18 years.
* Ability to understand and fill out questionnaires.
* Written informed consent.

Exclusion Criteria:

* Metastatic breast cancer (defined as secondary spread to other organs, such as bones, lung, liver, mediastinal lymph nodes) or DCIS.
* Other cancer diagnosis in the past 5 years except non-melanotic skin cancer or cervical intraepithelial neoplasia.
* Male breast cancer.
* Patients on maintenance therapy (other than endocrine therapy).
* Patients participating in interventional clinical studies with Quality of Life as primary endpoint.
* Any psychological (including preexisting psychiatric disorders), familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: EBC and LABC cancer patients after primary treatment attending participating hospitals for routine follow-up.
Sampling Method: Non-Probability Sample
Enrollment: 830 (Estimated)
Dates: Start 2020-10-14 (Actual); Primary Completion 2024-03-31 (Estimated); Study Completion 2024-04-30 (Estimated)

PRIMARY OUTCOMES:
Health-related quality of life | 18 months after first patient inclusion
  It will be evaluated using self-administered EORTC QLQ-C30 questionnaire
Health-related quality of life | 18 months after first patient inclusion
  It will be evaluated using self-administered EORTC-QLQ-BR-45 questionnaire
Health-related quality of life | 18 months after first patient inclusion
  It will be evaluated using self-administered EORTC OUT-PATSAT-C7 questionnaire
Health-related quality of life | 18 months after first patient inclusion
  It will be evaluated using self-administered EORTC Sexual Health Questionnaire
Health-related quality of life | 18 months after first patient inclusion
  It will be evaluated using self-administered Distress Thermometer

CONTACTS AND LOCATIONS:
Locations (28):
- Belgium (5):
  - Onze Lieve Vrouw Ziekenhuis, Aalst
  - CHU Saint Pierre - CHU Saint-Pierre-Site Porte de Hal, Brussels
  - Cliniques Universitaires Saint-Luc, Brussels
  - C.H.U. Sart-Tilman, Liège
  - CHU-UCL Namur - CHU Site Sainte-Elisabeth-UCL Namur, Namur
- France (2):
  - Assistance Publique Hopitaux Paris - Assistance Publique - Hopitaux de Paris - Hopital Tenon, Paris, De
  - Groupe Radiopole Artois - Centre de radiotherapie Marie Curie, Arras
- Germany (2):
  - Universitaetsklinikum Leipzig-Klinik fuer Strahlentherapie und Radioonkologie, Leipzig
  - HELIOS Kliniken - Helios Klinikum Wuppertal - Klin. Univ. Witten / Herdecke, Wuppertal
- Italy (6):
  - Ospedale Generale Regionale, Bolzano
  - Azienda Ospedaliero-Universitaria Careggi, Florence
  - Ospedale San Gerardo, Monza
  - IRCCS - Fondazione G. Pascale, Napoli
  - IRCCS - Istituto Oncologico Veneto, Padua
  - Universita Di Roma La Sapienza - Universita Degli Studi Di Roma La Sapienza - Ospedale Sant'Andrea, Roma
- King Hussein Cancer Center, Amman, Jordan
- The Netherlands Cancer Institute-Antoni Van Leeuwenhoekziekenhuis, Amsterdam, Netherlands
- Poland (3):
  - Medical University Of Gdansk, Gdansk
  - The Great Poland Cancer Centre, Poznan
  - Maria Sklodowska-Curie Memorial Cancer Centre - Maria Sklodowska-Curie National Research Institute of Oncology, Warsaw
- Spain (4):
  - Hospital Universitario Reina Sofia, Córdoba
  - Clinica Universidad de Navarra, Madrid
  - Hospital Universitario Ramon y Cajal, Madrid
  - Complejo Hospitalario de Navarra, Pamplona
- Switzerland (2):
  - Group Of Private Clinics Hirslanden - Hirslanden Klinik-Tumor Zentrum Aarau, Aarau
  - Tumor and Breast Center ZeTuP St. Gallen, Sankt Gallen
- United Kingdom (2):
  - Leeds Teaching Hospitals NHS Trust - St. James's University Hospital, Leeds
  - Barts Health NHS Trust - St. Bartholomew'S Hospital, London